CLINICAL TRIAL: NCT03197935
Title: A Phase III Randomized Study to Investigate the Efficacy and Safety of Atezolizumab (Anti-PD-L1 Antibody) in Combination With Neoadjuvant Anthracycline/Nab-Paclitaxel-Based Chemotherapy Compared With Placebo and Chemotherapy in Patients With Primary Invasive Triple-Negative Breast Cancer
Brief Title: A Study to Investigate Atezolizumab and Chemotherapy Compared With Placebo and Chemotherapy in the Neoadjuvant Setting in Participants With Early Stage Triple Negative Breast Cancer
Acronym: IMpassion031
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO39392; 2016-004734-22 (EudraCT Number)
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; 130-nm albumin-bound paclitaxel; Doxorubicin; Cyclophosphamide; Filgrastim; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab and Chemotherapy (Experimental): Participants received atezolizumab (840 milligrams [mg]) via intravenous (IV) infusion every 2 weeks in combination with nab-paclitaxel (125 milligrams per square meter [mg/m^2]) via IV infusion every week for 12 weeks, followed by atezolizumab (840 mg) every 2 weeks in combination with doxorubicin (60 mg/m^2) and cyclophosphamide (600 mg/m^2) every 2 weeks via IV infusions with filgrastim/pegfilgrastim support for 4 doses. Participants continued to receive unblinded atezolizumab post-surgery at a fixed dose of 1200 mg by IV infusion every 3 weeks for 11 doses, for a total of approximately 12 months of atezolizumab therapy.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PDL1 antibody; Drug: Nab-paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Filgrastim; Drug: Pegfilgrastim
- Placebo and Chemotherapy (Placebo Comparator): Participants received placebo matched to atezolizumab via IV infusion every 2 weeks in combination with nab-paclitaxel (125 mg/m^2) via IV infusion every week for 12 weeks, followed by placebo matched to atezolizumab every 2 weeks in combination with doxorubicin (60 mg/m^2) and cyclophosphamide (600 mg/m^2) every 2 weeks via IV infusions with filgrastim/pegfilgrastim support for 4 doses. Participants will be unblinded post-surgery and will continue to be followed.
  Interventions: Drug: Placebo; Drug: Nab-paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Filgrastim; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PDL1 antibody — Atezolizumab was administered as per schedule described in respective arm.
  Arms: Atezolizumab and Chemotherapy
Drug: Placebo — Placebo matched to atezolizumab was administered as per schedule described in respective arm.
  Arms: Placebo and Chemotherapy
Drug: Nab-paclitaxel — Nab-paclitaxel was administered as per schedule described in the arms.
Drug: Doxorubicin — Doxorubicin was administered as per schedule described in the arms.
Drug: Cyclophosphamide — Cyclophosphamide was administered as per schedule described in the arms.
Drug: Filgrastim — Filgrastim was administered according to local prescribing information as determined by the Investigator for 4 doses after completion of initial 12 weeks.
Drug: Pegfilgrastim — Pegfilgrastim was administered according to local prescribing information as determined by the Investigator for 4 doses after completion of initial 12 weeks.

SUMMARY:
This is a global Phase III, double-blind, randomized, placebo-controlled study designed to evaluate the efficacy and safety of neoadjuvant treatment with atezolizumab (anti-programmed death-ligand 1 [anti-PD-L1] antibody) and nab-paclitaxel followed by doxorubicin and cyclophosphamide (nab-pac-AC), or placebo and nab-pac-AC in participants eligible for surgery with initial clinically assessed triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically documented TNBC (negative human epidermal growth factor receptor 2 [HER2], estrogen receptor [ER], and progesterone receptor [PgR] status)
* Confirmed tumor programmed death-ligand 1 (PD-L1) evaluation as documented through central testing of a representative tumor tissue specimen
* Primary breast tumor size of greater than (>) 2 centimeters (cm) by at least one radiographic or clinical measurement
* Stage at presentation: cT2-cT4, cN0-cN3, cM0
* Participant agreement to undergo appropriate surgical management including axillary lymph node surgery and partial or total mastectomy after completion of neoadjuvant treatment
* Baseline left ventricular ejection fraction (LVEF) greater than or equal to (>=) 53 percent (%) measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scans
* Adequate hematologic and end-organ function
* Representative formalin-fixed, paraffin-embedded (FFPE) tumor specimen in paraffin blocks (preferred) or at least 20 unstained slides, with an associated pathology report documenting ER, PgR, and HER2 negativity
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm
* Women who are not postmenopausal or have undergone a sterilization procedure must have a negative serum pregnancy test result within 14 days prior to initiation of study drug

Exclusion criteria:

* Prior history of invasive breast cancer
* Stage 4 (metastatic) breast cancer
* Prior systemic therapy for treatment and prevention of breast cancer
* Previous therapy with anthracyclines or taxanes for any malignancy
* History of ductal carcinoma in situ (DCIS), except for participants treated exclusively with mastectomy >5 years prior to diagnosis of current breast cancer
* History of pleomorphic lobular carcinoma in situ (LCIS), except for participants surgically managed >5 years prior to diagnosis of current breast cancer
* Bilateral breast cancer
* Undergone incisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes
* Axillary lymph node dissection prior to initiation of neoadjuvant therapy
* History of other malignancy within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Cardiopulmonary dysfunction
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells
* Known allergy or hypersensitivity to the components of the formulations of atezolizumab, nab-paclitaxel, cyclophosphamide, or doxorubicin, filgrastim or pegfilgrastim
* Active or history of autoimmune disease or immune deficiency diseases except history of autoimmune-related hypothyroidism, controlled Type 1 diabetes mellitus, and dermatologic manifestations of eczema, psoriasis, lichen simplex chronicus, or vitiligo (e.g., participants with psoriatic arthritis are excluded)
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive human immunodeficiency virus (HIV) test at screening
* Active hepatitis B and hepatitis C virus infection
* Active tuberculosis
* Severe infections within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment, except prophylactic antibiotics
* Major surgical procedure within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study
* Prior allogeneic stem cell or solid organ transplantation
* Administration of a live attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint-blockade therapies, including anti-cluster of differentiation 40 (anti-CD40), anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to initiation of study treatment
* Treatment with systemic immunosuppressive medications within 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressive medications during the study
* History of cerebrovascular accident within 12 months prior to randomization
* Pregnant or lactating, or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (68):
- United States (12):
  - Stanford University Medical Center, Palo Alto, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Carrollton, Georgia
  - Mercy Medical Center, Baltimore, Maryland
  - HCA Midwest Division, Kansas City, Missouri
  - The Valley Hospital; Valley Medical Group, Paramus, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology - Chattanooga; Tennessee Oncology - East Third Street, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - Cancer Care Northwest, Spokane, Washington
- Australia (2):
  - Monash Medical Centre, Clayton, Victoria
  - Fiona Stanley Hospital; FSH Cancer Centre Clinical Trials Unit, Bull Creek, Western Australia
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Ste-Elisabeth, Namur
  - Sint Augustinus Wilrijk, Wilrijk
- Brazil (8):
  - Santa Casa de Misericordia de Salvador, Salvador, Estado de Bahia
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - CETUS Hospital Dia Oncologia, Uberaba, Minas Gerais
  - Iop Instituto de Oncologia Do Parana, Curitiba, Paraná
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- Canada (3):
  - Jewish General Hospital, Montreal, Quebec
  - Hopital Sacre-Coeur Research Centre, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- Germany (13):
  - Hochwaldkrankenhaus, Bad Nauheim
  - Praxisklinik Krebsheilkunde für Frauen / Brustzentrum (Dres. Kittel/Klare), Berlin
  - Ambulantes Tumorzentrum Spandau; Dres. Benno Mohr und Uwe Peters, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Luisenkrankenhaus GmbH & Co. KG., Brustzentrum, Düsseldorf
  - Evangelische Kliniken Gelsenkirchen GmbH; Brustzentrum, Gelsenkirchen
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - Diakovere Henriettenstift, Frauenklinik, Hanover
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - St. Elisabeth-Krankenhaus, Senologie/Brustzentrum, Leipzig
  - Klinik & Poliklinik für Frauenheilkunde und Geburtshilfe, Campus Innenstadt, München
  - Universitätsklinikum Münster; Klinik für Frauenheilkunde und Geburtshilfe, Münster
  - Medizinisches Versorgungszentrum am Klinikum Oldenburg GmbH, Oldenburg
- Italy (3):
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - Azienda ULSS 8 Berica; Oncologia Medica - Ospedlae di Vicenza, Vicenza, Veneto
- Japan (9):
  - Aichi Cancer Center Hospital, Aichi
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - Fukushima Medical University Hospital, Fukushima
  - Hiroshima City Hiroshima Citizens Hospital; Breast Surgery, Hiroshima
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - National Hospital Organization Osaka National Hospital; Breast Surgery, Osaka
  - St. Luke's Internat. Hospital, Breast Surgical Oncology, Tokyo
  - The Cancer Inst. Hosp. of JFCR; Breast Oncology Center, Tokyo
- Poland (2):
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad; Klinika Nowtw.Piersi i Chir.Rekonstr, Warsaw
  - Dolnoslaskie Centrum Onkologii, Pulmonologii i Hematologii; Oddz. Onkologii Klin. i Chemioterapii, Wroc?aw
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
- Taiwan (3):
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - Mackay Memorial Hospital; Dept of Surgery, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester
  - Barts & London School of Med; Medical Oncology, London
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Mittendorf EA, Assaf ZJ, Harbeck N, Zhang H, Saji S, Jung KH, Hegg R, Koehler A, Sohn J, Iwata H, Telli ML, Ferrario C, Punie K, Qamra A, Dieterich M, Xu Y, Liste-Hermoso M, Shearer-Kang E, Molinero L, Chui SY, Barrios CH. Peri-operative atezolizumab in early-stage triple-negative breast cancer: final results and ctDNA analyses from the randomized phase 3 IMpassion031 trial. Nat Med. 2025 Jul;31(7):2397-2404. doi: 10.1038/s41591-025-03725-4. Epub 2025 Jun 4. PMID 40467898
- [Derived] Mittendorf EA, Zhang H, Barrios CH, Saji S, Jung KH, Hegg R, Koehler A, Sohn J, Iwata H, Telli ML, Ferrario C, Punie K, Penault-Llorca F, Patel S, Duc AN, Liste-Hermoso M, Maiya V, Molinero L, Chui SY, Harbeck N. Neoadjuvant atezolizumab in combination with sequential nab-paclitaxel and anthracycline-based chemotherapy versus placebo and chemotherapy in patients with early-stage triple-negative breast cancer (IMpassion031): a randomised, double-blind, phase 3 trial. Lancet. 2020 Oct 10;396(10257):1090-1100. doi: 10.1016/S0140-6736(20)31953-X. Epub 2020 Sep 20. PMID 32966830
- [Derived] Perez-Garcia J, Soberino J, Racca F, Gion M, Stradella A, Cortes J. Atezolizumab in the treatment of metastatic triple-negative breast cancer. Expert Opin Biol Ther. 2020 Sep;20(9):981-989. doi: 10.1080/14712598.2020.1769063. Epub 2020 May 25. PMID 32450725

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo and Chemotherapy: Participants received placebo matched to atezolizumab via IV infusion every 2 weeks in combination with nab-paclitaxel (125 mg/m^2) via IV infusion every week for 12 weeks, followed by placebo matched to atezolizumab every 2 weeks in combination with doxorubicin (60 mg/m^2) and cyclophosphamide (600 mg/m^2) every 2 weeks via IV infusions with filgrastim/pegfilgrastim support for 4 doses. Participants will continue to be followed after surgery.
Period: Overall Study
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Started | 168 | 165
Completed | 121 | 136
Not Completed | 47 | 29
Not completed — Death due to any cause | 26 | 15
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 16 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy | Total
Number analyzed (Participants) | 168 | 165 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (13.2) | 50.1 (11.6) | 50.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 165 | 333
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 45 | 92
  Not Hispanic or Latino | 114 | 114 | 228
  Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 41 | 47 | 88
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 9 | 24
  White | 108 | 102 | 210
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR) Using American Joint Committee on Cancer (AJCC) Staging System in ITT Population
Description: Number of participants with Pathologic Complete Response (pCR) Using American Joint Committee on Cancer (AJCC) Staging System in ITT Population. pCR is defined as eradication of invasive tumor from both breast and lymph nodes (ypT0/is ypN0). pCR was evaluated for each participant after neoadjuvant study treatment and surgery. Participants whose pCR assessment was missing will be counted as not achieving a pCR.
Time Frame: After neoadjuvant study treatment and surgery, up to primary analysis data cut off on 03 ApriI 2020
Population: ITT population (full population) is defined as all randomized participants.
Measure: Number; unit: Number of Participants
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 168 | 165
Number of Participants | 69 | 95
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: tumor PD-L1 status (IC0 vs. IC1/2/3) and clinical stage at presentation (Stage II vs. III); Test type: Superiority; p = 0.0044, Cochran-Mantel-Haenszel — (one-sided); Absolute difference in pCR rate = 16.50, 95% CI 2-sided [5.91 to 27.10]

2. Primary Outcome: Number of Participants With pCR in Subpopulation With PD-L1-Positive Tumor Status (Tumor-infiltrating Immune Cell [IC] 1/2/3) Using AJCC Staging System
Description: Number of participants with Pathologic Complete Response (pCR) Using American Joint Committee on Cancer (AJCC) Staging System in the subpopulation with programmed death-ligand1 (PD-L1)-positive tumor status(tumor-infiltrating immune cell [IC] IC1/2/3) . pCR is defined as eradication of invasive tumor from both breast and lymph nodes (ypT0/is ypN0). pCR was evaluated for each participant after neoadjuvant study treatment and surgery. Participants whose pCR assessment was missing will be counted as not achieving a pCR.
Time Frame: After neoadjuvant study treatment and surgery, up to primary analysis data cut off on 03 ApriI 2020
Population: PD-L1-positive subpopulation is defined as participants in the ITT population whose PD-L1 status is IC1/2/3 at the time of randomization.
Measure: Number; unit: Number of Participants
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 75 | 77
Number of Participants | 37 | 53
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: AJCC stage at diagnosis (II vs. III); Test type: Superiority; p = 0.0206, Cochran-Mantel-Haenszel — (one-sided); Difference in pCR = 19.50, 95% CI 2-sided [4.17 to 34.83]

3. Secondary Outcome: Event-Free Survival (EFS) in All Participants
Description: Event-free survival (EFS) defined as the time from randomization to the first documented occurrence of disease recurrence, disease progression, or death from any cause in all participants. Recurrent disease includes local, regional, or distant recurrence and contralateral breast cancer. Ipsilateral or contralateral in situ disease and second primary non-breast cancers (including in situ carcinomas and non-melanoma skin cancers) will not be counted as progressive disease or recurrent disease.
Time Frame: From randomization and up to study final analysis data cut off on 28 September 2022.
Population: ITT population (full population) is defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 168 | 165
Months | NA [NA to NA] — Not estimable due low number of events. | NA [NA to NA] — Not estimable due low number of events.
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: Tumor PD-L1 status (IC0 vs IC1/2/3) and AJCC stage at diagnosis (II vs. III); Test type: Other — This study was not designed nor formally powered to demonstrate statistically significant improvements in the secondary efficacy endpoint of EFS. The analyses of this secondary endpoint is descriptive in nature; Stratified log-rank test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.47 to 1.21]

4. Secondary Outcome: Event-Free Survival (EFS) in Subpopulation With PD-L1-Postive Tumor Status
Description: Event-free survival (EFS) defined as the time from randomization to the first documented occurrence of disease recurrence, disease progression, or death from any cause in the subpopulation with PD-L1-positive tumor status. Recurrent disease includes local, regional, or distant recurrence and contralateral breast cancer. Ipsilateral or contralateral in situ disease and second primary non-breast cancers (including in situ carcinomas and non-melanoma skin cancers) will not be counted as progressive disease or recurrent disease.
Time Frame: From randomization and up to study final analysis data cut off on 28 September 2022.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 75 | 77
Months | NA [NA to NA] — Not estimable due low number of events. | NA [NA to NA] — Not estimable due low number of events.
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: AJCC stage at diagnosis (II vs. III); Test type: Other — [test comment as in outcome 3, analysis 1]; Stratified log-rank test; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.26 to 1.18]

5. Secondary Outcome: Disease-Free Survival (DFS) in All Participants Who Undergo Surgery
Description: Disease-free survival (DFS) defined as the time from surgery to the first documented disease recurrence or death from any cause, whichever occurs first. DFS is analyzed with the use of the same methodology as specified for EFS for all participants.
Time Frame: From surgery and up to study final analysis data cut off on 28 September 2022.
Population: ITT population (full population) is defined as all randomized participants. Participants who do not undergo surgery at the end of neoadjuvant treatment are excluded from the analysis of DFS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 153 | 155
Months | NA [NA to NA] — Not estimable due low number of events. | NA [NA to NA] — Not estimable due low number of events.
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: Tumor PD-L1 status (IC0 vs IC1/2/3) and AJCC stage at diagnosis (II vs. III); Test type: Other — This study was not designed nor formally powered to demonstrate statistically significant improvements in the secondary efficacy endpoint of DFS. The analyses of this secondary endpoint are descriptive in nature; Stratified log-rank test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.44 to 1.30]

6. Secondary Outcome: Disease-Free Survival (DFS) in Subpopulation of Participants With PD-L1-Positive Tumor Status Who Undergo Surgery
Description: Disease-free survival (DFS) defined as the time from surgery to the first documented disease recurrence or death from any cause, whichever occurs first. DFS is analyzed with the use of the same methodology as specified for EFS for the subpopulation of participants with PD-L1-positive tumor status.
Time Frame: From surgery and up to study final analysis data cut off on 28 September 2022.
Population: PD-L1-positive subpopulation is defined as participants in the ITT population whose PD-L1 status is IC1/2/3 at the time of randomization. Participants who do not undergo surgery at the end of neoadjuvant treatment are excluded from the analysis of DFS in the Subpopulation of Participants with PD-L1-Positive Tumor Status.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 67 | 73
Months | NA [NA to NA] — Not estimable due low number of events. | NA [NA to NA] — Not estimable due low number of events.
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: AJCC stage at diagnosis (II vs. III); Test type: Other — [test comment as in outcome 5, analysis 1]; Stratified log-rank test; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.23 to 1.43]

7. Secondary Outcome: Overall Survival (OS) in All Participants
Description: Overall survival (OS) defined as the time from randomization to the date of death from any cause in all participants.
Time Frame: From randomization and up to study final analysis data cut off on 28 September 2022.
Population: ITT population (full population) is defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 168 | 165
Months | NA [NA to NA] — Not estimable due low number of events. | NA [NA to NA] — Not estimable due low number of events.
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: Tumor PD-L1 status (IC0 vs IC1/2/3) and AJCC stage at diagnosis (II vs. III); Test type: Other — This study was not designed nor formally powered to demonstrate statistically significant improvements in the secondary efficacy endpoints of OS. The analyses of this secondary endpoint are descriptive in nature; Stratified log-rank test; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.30 to 1.04]

8. Secondary Outcome: Overall Survival (OS) in Subpopulation With PD-L1-Positive Tumor Status
Description: Overall survival (OS) defined as the time from randomization to the date of death from any cause in the subpopulation with PD-L1-positive tumor status.
Time Frame: From randomization and up to study final analysis data cut off on 28 September 2022.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 75 | 77
Months | NA [NA to NA] — Not estimable due low number of events. | NA [NA to NA] — Not estimable due low number of events.
Statistical Analysis 1: Comparison: Placebo and Chemotherapy vs Atezolizumab and Chemotherapy; Stratified analysis. Strata are: AJCC stage at diagnosis (II vs. III); Test type: Other — This study was not designed nor formally powered to demonstrate statistically significant improvements in the secondary efficacy endpoints of EFS, DFS and OS. The analyses of this secondary endpoint are descriptive in nature; Stratified log-rank test; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.26 to 1.91]

9. Secondary Outcome: Mean Scores for Function (Role/Physical) and GHS/HRQoL by Cycle and Between Treatment Arms as Assessed by the EORTC QLQ-C30
Description: Mean score in function (role, physical) and global health status(GHS)/ health-related quality of life (HRQoL) by cycle and between treatment arms as assessed by the functional and HRQoL scales of the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core30(QLQ C30). The score range for each scale and single-item measure is 0 to 100, where higher scores indicate a higher response level (i.e., better functioning, better QoL, worse symptoms).
Time Frame: From randomization and up to study final analysis data cut off on 28 September 2022.
Population: All randomized participants with non-missing baseline assessment and at least one non-missing post-baseline assessment.
Measure: Mean (95% Confidence Interval); unit: Score on a 0-100 scale
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 167 | 161
Score on a 0-100 scale
  GHS/QoL Baseline | 76.45 [73.47 to 79.42] | 79.24 [76.34 to 82.14]
  GHS/QoL Cycle 2 Day 1: number analyzed (Participants) | 164 | 157
  GHS/QoL Cycle 2 Day 1 | 71.90 [69.04 to 74.76] | 71.55 [68.53 to 74.57]
  GHS/QoL Cycle 3 Day 1: number analyzed (Participants) | 152 | 143
  GHS/QoL Cycle 3 Day 1 | 65.30 [62.25 to 68.34] | 62.65 [58.94 to 66.36]
  GHS/QoL Cycle 4 Day 1: number analyzed (Participants) | 153 | 149
  GHS/QoL Cycle 4 Day 1 | 62.36 [59.15 to 65.58] | 59.84 [56.62 to 63.07]
  GHS/QoL Cycle Cycle 5 Day 1: number analyzed (Participants) | 147 | 139
  GHS/QoL Cycle Cycle 5 Day 1 | 60.37 [56.87 to 63.87] | 53.60 [49.71 to 57.48]
  GHS/QoL Cycle 6 Day 1: number analyzed (Participants) | 134 | 132
  GHS/QoL Cycle 6 Day 1 | 74.25 [70.86 to 77.65] | 70.14 [66.97 to 73.31]
  GHS/QoL Cycle 7 Day 1: number analyzed (Participants) | 122 | 128
  GHS/QoL Cycle 7 Day 1 | 76.50 [73.39 to 79.62] | 73.57 [70.92 to 76.22]
  GHS/QoL Cycle 8 Day 1: number analyzed (Participants) | 119 | 122
  GHS/QoL Cycle 8 Day 1 | 77.17 [74.35 to 79.99] | 72.06 [69.01 to 75.11]
  GHS/QoL Cycle 9 Day 1: number analyzed (Participants) | 121 | 121
  GHS/QoL Cycle 9 Day 1 | 75.62 [72.54 to 78.69] | 72.18 [69.18 to 75.17]
  GHS/QoL Cycle 10 Day 1: number analyzed (Participants) | 114 | 122
  GHS/QoL Cycle 10 Day 1 | 75.22 [72.22 to 78.22] | 70.56 [67.09 to 74.03]
  GHS/QoL Cycle 11 Day 1: number analyzed (Participants) | 119 | 122
  GHS/QoL Cycle 11 Day 1 | 75.98 [73.17 to 78.79] | 71.93 [68.53 to 75.32]
  GHS/QoL Cycle 12 Day 1: number analyzed (Participants) | 119 | 122
  GHS/QoL Cycle 12 Day 1 | 75.84 [72.93 to 78.75] | 72.40 [69.27 to 75.54]
  GHS/QoL Cycle 13 Day 1: number analyzed (Participants) | 119 | 121
  GHS/QoL Cycle 13 Day 1 | 74.72 [71.35 to 78.08] | 72.87 [69.67 to 76.06]
  GHS/QoL Cycle 14 Day 1: number analyzed (Participants) | 119 | 116
  GHS/QoL Cycle 14 Day 1 | 74.79 [71.61 to 77.97] | 71.19 [67.65 to 74.43]
  GHS/QoL Cycle 15 Day 1: number analyzed (Participants) | 112 | 116
  GHS/QoL Cycle 15 Day 1 | 75.00 [71.85 to 78.15] | 74.07 [71.08 to 77.06]
  GHS/QoL Cycle 16 Day 1: number analyzed (Participants) | 111 | 114
  GHS/QoL Cycle 16 Day 1 | 77.70 [74.70 to 80.71] | 74.93 [71.69 to 78.16]
  GHS/QoL Study Drug Completion/ Early Discontinuation: number analyzed (Participants) | 130 | 137
  GHS/QoL Study Drug Completion/ Early Discontinuation | 75.38 [72.18 to 78.59] | 72.51 [68.96 to 76.05]
  GHS/QoL Survival Follow-Up Month 3: number analyzed (Participants) | 131 | 142
  GHS/QoL Survival Follow-Up Month 3 | 76.97 [73.87 to 80.07] | 72.65 [69.33 to 75.98]
  GHS/QoL Survival Follow-Up Month 6: number analyzed (Participants) | 125 | 136
  GHS/QoL Survival Follow-Up Month 6 | 74.93 [71.28 to 78.59] | 75.61 [72.09 to 79.14]
  GHS/QoL Survival Follow-Up Month 9: number analyzed (Participants) | 116 | 132
  GHS/QoL Survival Follow-Up Month 9 | 75.00 [71.32 to 76.68] | 75.19 [71.78 to 78.60]
  GHS/QoL Survival Follow-Up Month 12: number analyzed (Participants) | 111 | 126
  GHS/QoL Survival Follow-Up Month 12 | 75.15 [71.66 to 78.64] | 74.87 [71.13 to 78.60]
  GHS/QoL Survival Follow-Up Month 18: number analyzed (Participants) | 102 | 112
  GHS/QoL Survival Follow-Up Month 18 | 76.39 [72.29 to 80.48] | 75.60 [72.01 to 79.18]
  GHS/QoL Survival Follow-Up Month 24: number analyzed (Participants) | 83 | 108
  GHS/QoL Survival Follow-Up Month 24 | 78.31 [74.89 to 81.73] | 74.46 [70.55 to 78.37]
  GHS/QoL Survival Follow-Up Month 30: number analyzed (Participants) | 65 | 72
  GHS/QoL Survival Follow-Up Month 30 | 78.33 [74.08 to 82.59] | 73.50 [68.56 to 78.43]
  GHS/QoL Survival Follow-Up Month 36: number analyzed (Participants) | 62 | 69
  GHS/QoL Survival Follow-Up Month 36 | 78.63 [74.53 to 82.73] | 76.93 [71.85 to 82.01]
  GHS/QoL Survival Follow-Up Month 48: number analyzed (Participants) | 2 | 7
  GHS/QoL Survival Follow-Up Month 48 | 58.33 [-259.32 to 375.99] | 63.10 [47.77 to 78.42]
  Physical Functioning Baseline: number analyzed (Participants) | 166 | 161
  Physical Functioning Baseline | 90.03 [87.82 to 92.24] | 90.85 [88.53 to 93.17]
  Physical Functioning Cycle 2 Day 1: number analyzed (Participants) | 164 | 157
  Physical Functioning Cycle 2 Day 1 | 83.50 [80.79 to 86.21] | 84.93 [82.55 to 87.31]
  Physical Functioning Cycle 3 Day 1: number analyzed (Participants) | 152 | 142
  Physical Functioning Cycle 3 Day 1 | 78.33 [75.19 to 81.48] | 77.29 [74.04 to 80.54]
  Physical Functioning Cycle 4 Day 1: number analyzed (Participants) | 152 | 149
  Physical Functioning Cycle 4 Day 1 | 70.42 [67.06 to 73.77] | 69.02 [65.52 to 72.51]
  Physical Functioning Cycle 5 Day 1: number analyzed (Participants) | 146 | 139
  Physical Functioning Cycle 5 Day 1 | 67.91 [64.18 to 71.65] | 64.27 [60.40 to 68.13]
  Physical Functioning Cycle 6 Day 1: number analyzed (Participants) | 134 | 132
  Physical Functioning Cycle 6 Day 1 | 79.49 [76.38 to 82.60] | 78.01 [74.81 to 81.20]
  Physical Functioning Cycle 7 Day 1: number analyzed (Participants) | 122 | 128
  Physical Functioning Cycle 7 Day 1 | 82.73 [79.76 to 85.71] | 80.78 [77.96 to 83.60]
  Physical Functioning Cycle 8 Day 1: number analyzed (Participants) | 119 | 122
  Physical Functioning Cycle 8 Day 1 | 85.15 [82.75 to 87.56] | 81.75 [78.59 to 84.90]
  Physical Functioning Cycle 9 Day 1: number analyzed (Participants) | 121 | 122
  Physical Functioning Cycle 9 Day 1 | 84.19 [81.57 to 86.81] | 83.99 [81.36 to 86.62]
  Physical Functioning Cycle 10 Day 1: number analyzed (Participants) | 114 | 122
  Physical Functioning Cycle 10 Day 1 | 84.78 [82.16 to 87.40] | 83.88 [81.21 to 86.55]
  Physical Functioning Cycle 11 Day 1: number analyzed (Participants) | 119 | 121
  Physical Functioning Cycle 11 Day 1 | 85.48 [83.18 to 87.77] | 84.24 [81.33 to 87.15]
  Physical Functioning Cycle 12 Day 1: number analyzed (Participants) | 119 | 122
  Physical Functioning Cycle 12 Day 1 | 86.97 [84.66 to 89.29] | 83.44 [80.55 to 86.34]
  Physical Functioning Cycle 13 Day 1: number analyzed (Participants) | 119 | 121
  Physical Functioning Cycle 13 Day 1 | 86.16 [83.40 to 88.93] | 83.36 [80.27 to 86.45]
  Physical Functioning Cycle 14 Day 1: number analyzed (Participants) | 119 | 117
  Physical Functioning Cycle 14 Day 1 | 86.22 [83.56 to 88.88] | 84.96 [82.18 to 87.73]
  Physical Functioning Cycle 15 Day 1: number analyzed (Participants) | 112 | 116
  Physical Functioning Cycle 15 Day 1 | 84.69 [81.67 to 87.71] | 84.28 [81.23 to 87.34]
  Physical Functioning Cycle 16 Day 1: number analyzed (Participants) | 111 | 114
  Physical Functioning Cycle 16 Day 1 | 87.19 [84.34 to 90.04] | 84.33 [81.37 to 87.29]
  Physical Functioning Drug Completion/Early Discontinuation: number analyzed (Participants) | 130 | 137
  Physical Functioning Drug Completion/Early Discontinuation | 84.21 [81.31 to 87.10] | 82.34 [79.24 to 85.43]
  Physical Functioning Survival Follow-Up Month 3: number analyzed (Participants) | 131 | 142
  Physical Functioning Survival Follow-Up Month 3 | 85.29 [82.65 to 87.93] | 82.35 [79.29 to 85.41]
  Physical Functioning Survival Follow-Up Month 6: number analyzed (Participants) | 125 | 136
  Physical Functioning Survival Follow-Up Month 6 | 84.96 [82.15 to 87.77] | 84.17 [81.11 to 87.22]
  Physical Functioning Survival Follow-Up Month 9: number analyzed (Participants) | 116 | 132
  Physical Functioning Survival Follow-Up Month 9 | 85.11 [82.46 to 87.77] | 83.48 [80.01 to 86.96]
  Physical Functioning Survival Follow-Up Month 12: number analyzed (Participants) | 111 | 126
  Physical Functioning Survival Follow-Up Month 12 | 85.05 [81.79 to 88.30] | 83.17 [79.67 to 86.68]
  Physical Functioning Survival Follow-Up Month 18: number analyzed (Participants) | 102 | 112
  Physical Functioning Survival Follow-Up Month 18 | 85.23 [81.63 to 88.82] | 84.29 [80.85 to 87.72]
  Physical Functioning Survival Follow-Up Month 24: number analyzed (Participants) | 82 | 108
  Physical Functioning Survival Follow-Up Month 24 | 85.69 [82.05 to 89.33] | 85.43 [81.67 to 89.20]
  Physical Functioning Survival Follow-Up Month 30: number analyzed (Participants) | 65 | 72
  Physical Functioning Survival Follow-Up Month 30 | 87.08 [83.41 to 90.75] | 84.54 [80.35 to 88.73]
  Physical Functioning Survival Follow-Up Month 36: number analyzed (Participants) | 62 | 69
  Physical Functioning Survival Follow-Up Month 36 | 86.24 [81.63 to 90.84] | 85.80 [81.87 to 89.73]
  Physical Functioning Survival Follow-Up Month 48: number analyzed (Participants) | 2 | 7
  Physical Functioning Survival Follow-Up Month 48 | 90.00 [-37.06 to 217.06] | 88.57 [75.88 to 101.26]
  Role Functioning Baseline: number analyzed (Participants) | 166 | 161
  Role Functioning Baseline | 88.86 [85.67 to 92.04] | 89.44 [86.10 to 92.78]
  Role Functioning Cycle 2 Day 1: number analyzed (Participants) | 164 | 157
  Role Functioning Cycle 2 Day 1 | 80.39 [76.77 to 84.00] | 77.18 [73.47 to 80.88]
  Role Functioning Cycle 3 Day 1: number analyzed (Participants) | 152 | 142
  Role Functioning Cycle 3 Day 1 | 70.39 [65.96 to 74.83] | 69.48 [65.29 to 73.67]
  Role Functioning Cycle 4 Day 1: number analyzed (Participants) | 153 | 149
  Role Functioning Cycle 4 Day 1 | 61.11 [56.70 to 65.53] | 56.60 [51.56 to 61.64]
  Role Functioning Cycle 5 Day 1: number analyzed (Participants) | 146 | 139
  Role Functioning Cycle 5 Day 1 | 56.06 [51.06 to 61.04] | 51.08 [46.15 to 56.00]
  Role Functioning Cycle 6 Day 1: number analyzed (Participants) | 134 | 132
  Role Functioning Cycle 6 Day 1 | 66.17 [61.45 to 70.89] | 62.88 [57.70 to 68.06]
  Role Functioning Cycle 7 Day 1: number analyzed (Participants) | 122 | 128
  Role Functioning Cycle 7 Day 1 | 73.77 [69.21 to 78.33] | 69.92 [65.46 to 74.39]
  Role Functioning Cycle 8 Day 1: number analyzed (Participants) | 119 | 122
  Role Functioning Cycle 8 Day 1 | 77.59 [73.57 to 81.62] | 72.95 [68.13 to 77.77]
  Role Functioning Cycle 9 Day 1: number analyzed (Participants) | 121 | 122
  Role Functioning Cycle 9 Day 1 | 77.13 [72.98 to 81.29] | 74.32 [70.21 to 78.42]
  Role Functioning Cycle 10 Day 1: number analyzed (Participants) | 114 | 122
  Role Functioning Cycle 10 Day 1 | 78.51 [74.50 to 82.51] | 75.27 [70.94 to 79.61]
  Role Functioning Cycle 11 Day 1: number analyzed (Participants) | 119 | 122
  Role Functioning Cycle 11 Day 1 | 79.97 [76.41 to 83.53] | 75.68 [71.44 to 79.93]
  Role Functioning Cycle 12 Day 1: number analyzed (Participants) | 119 | 122
  Role Functioning Cycle 12 Day 1 | 81.79 [78.04 to 85.55] | 75.14 [70.52 to 79.75]
  Role Functioning Cycle 13 Day 1: number analyzed (Participants) | 119 | 121
  Role Functioning Cycle 13 Day 1 | 81.79 [78.16 to 85.42] | 74.38 [69.60 to 79.16]
  Role Functioning Cycle 14 Day 1: number analyzed (Participants) | 119 | 117
  Role Functioning Cycle 14 Day 1 | 80.81 [76.61 to 85.01] | 75.50 [70.60 to 80.40]
  Role Functioning Cycle 15 Day 1: number analyzed (Participants) | 112 | 116
  Role Functioning Cycle 15 Day 1 | 79.02 [75.14 to 82.90] | 77.59 [73.05 to 82.13]
  Role Functioning Cycle 16 Day 1: number analyzed (Participants) | 111 | 114
  Role Functioning Cycle 16 Day 1 | 83.03 [78.87 to 87.20] | 78.65 [74.05 to 83.26]
  Role Functioning Study Drug Completion/Early Discontinuation: number analyzed (Participants) | 130 | 137
  Role Functioning Study Drug Completion/Early Discontinuation | 80.00 [76.07 to 83.93] | 74.09 [69.37 to 78.81]
  Role Functioning Survival Follow-Up Month 3: number analyzed (Participants) | 131 | 142
  Role Functioning Survival Follow-Up Month 3 | 81.93 [78.24 to 85.63] | 75.47 [70.97 to 79.97]
  Role Functioning Survival Follow-Up Month 6: number analyzed (Participants) | 126 | 136
  Role Functioning Survival Follow-Up Month 6 | 78.53 [74.01 to 83.06] | 76.10 [71.38 to 80.83]
  Role Functioning Survival Follow-Up Month 9: number analyzed (Participants) | 116 | 132
  Role Functioning Survival Follow-Up Month 9 | 81.61 [77.90 to 85.32] | 76.39 [71.36 to 81.42]
  Role Functioning Survival Follow-Up Month 12: number analyzed (Participants) | 111 | 126
  Role Functioning Survival Follow-Up Month 12 | 81.68 [77.46 to 85.91] | 76.98 [71.47 to 82.50]
  Role Functioning Survival Follow-Up Month 18: number analyzed (Participants) | 102 | 112
  Role Functioning Survival Follow-Up Month 18 | 81.86 [76.88 to 86.85] | 77.98 [72.77 to 83.18]
  Role Functioning Survival Follow-Up Month 24: number analyzed (Participants) | 82 | 108
  Role Functioning Survival Follow-Up Month 24 | 79.47 [73.62 to 85.32] | 80.09 [75.03 to 85.15]
  Role Functioning Survival Follow-Up Month 30: number analyzed (Participants) | 65 | 72
  Role Functioning Survival Follow-Up Month 30 | 81.54 [75.51 to 87.56] | 78.24 [71.20 to 85.28]
  Role Functioning Survival Follow-Up Month 36: number analyzed (Participants) | 62 | 69
  Role Functioning Survival Follow-Up Month 36 | 85.48 [79.88 to 91.09] | 81.64 [75.23 to 88.05]
  Role Functioning Survival Follow-Up Month 48: number analyzed (Participants) | 2 | 7
  Role Functioning Survival Follow-Up Month 48 | 83.33 [-128.44 to 295.10] | 76.19 [-228.44 to 195.10]

10. Secondary Outcome: Mean Change From Baseline Scores for Function (Role, Physical) and GHS/HRQoL by Cycle and Between Treatment Arms as Assessed by the EORTC QLQ-C30
Description: Mean change from baseline score in function (role, physical) and global health status(GHS)/ health-related quality of life (HRQoL) by cycle and between treatment arms as assessed by the functional and HRQoL scales of the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core30(QLQ C30).
Time Frame: From randomization and up to study final analysis data cut off on 28 September 2022.
Population: All randomized participants with non-missing baseline assessment and at least one non-missing post-baseline assessment.
Measure: Mean (95% Confidence Interval); unit: Score on a 0-100 scale.
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 167 | 161
Score on a 0-100 scale.
  GHS/QoL Cycle 2 Day 1: number analyzed (Participants) | 164 | 157
  GHS/QoL Cycle 2 Day 1 | -4.62 [-7.89 to -1.36] | -7.91 [-11.09 to -4.72]
  GHS/QoL Cycle 3 Day 1: number analyzed (Participants) | 152 | 143
  GHS/QoL Cycle 3 Day 1 | -12.72 [-16.34 to -9.10] | -17.07 [-21.15 to -13.00]
  GHS/QoL Cycle 4 Day 1: number analyzed (Participants) | 153 | 149
  GHS/QoL Cycle 4 Day 1 | -14.49 [-18.35 to -10.62] | -19.80 [-23.50 to -16.09]
  GHS/QoL Cycle Cycle 5 Day 1: number analyzed (Participants) | 147 | 139
  GHS/QoL Cycle Cycle 5 Day 1 | -17.06 [-21.18 to -12.94] | -26.02 [-30.34 to -21.70]
  GHS/QoL Cycle 6 Day 1: number analyzed (Participants) | 134 | 132
  GHS/QoL Cycle 6 Day 1 | -2.49 [-6.70 to 1.72] | -8.78 [-12.71 to -4.84]
  GHS/QoL Cycle 7 Day 1: number analyzed (Participants) | 122 | 128
  GHS/QoL Cycle 7 Day 1 | -0.61 [-4.64 to 3.41] | -5.40 [-9.15 to -1.66]
  GHS/QoL Cycle 8 Day 1: number analyzed (Participants) | 119 | 122
  GHS/QoL Cycle 8 Day 1 | 0.77 [-3.30 to 4.84] | -6.69 [-10.49 to -2.90]
  GHS/QoL Cycle 9 Day 1: number analyzed (Participants) | 121 | 121
  GHS/QoL Cycle 9 Day 1 | -0.28 [-4.10 to 3.55] | -6.13 [-9.94 to -2.32]
  GHS/QoL Cycle 10 Day 1: number analyzed (Participants) | 114 | 122
  GHS/QoL Cycle 10 Day 1 | -1.17 [-5.02 to 2.68] | -8.40 [-12.50 to -4.30]
  GHS/QoL Cycle 11 Day 1: number analyzed (Participants) | 119 | 122
  GHS/QoL Cycle 11 Day 1 | 0.35 [-3.42 to 4.13] | -7.04 [-11.11 to -2.96]
  GHS/QoL Cycle 12 Day 1: number analyzed (Participants) | 119 | 122
  GHS/QoL Cycle 12 Day 1 | -0.63 [-4.64 to 3.38] | -6.56 [-10.48 to -2.64]
  GHS/QoL Cycle 13 Day 1: number analyzed (Participants) | 119 | 121
  GHS/QoL Cycle 13 Day 1 | -1.26 [-5.19 to 2.67] | -5.85 [-9.83 to -1.88]
  GHS/QoL Cycle 14 Day 1: number analyzed (Participants) | 119 | 116
  GHS/QoL Cycle 14 Day 1 | -1.05 [-4.95 to 2.85] | -7.47 [-11.44 to -3.50]
  GHS/QoL Cycle 15 Day 1: number analyzed (Participants) | 112 | 116
  GHS/QoL Cycle 15 Day 1 | 0.00 [-4.21 to 4.21] | -4.67 [-8.71 to -0.63]
  GHS/QoL Cycle 16 Day 1: number analyzed (Participants) | 111 | 114
  GHS/QoL Cycle 16 Day 1 | 2.10 [-1.66 to 5.86] | -3.73 [-7.93 to 0.48]
  GHS/QoL Study Drug Completion/ Early Discontinuation: number analyzed (Participants) | 130 | 137
  GHS/QoL Study Drug Completion/ Early Discontinuation | 0.06 [-3.99 to 4.12] | -6.20 [-10.47 to -1.94]
  GHS/QoL Survival Follow-Up Month 3: number analyzed (Participants) | 131 | 142
  GHS/QoL Survival Follow-Up Month 3 | 0.64 [-3.54 to 4.81] | -6.57 [-10.28 to -2.87]
  GHS/QoL Survival Follow-Up Month 6: number analyzed (Participants) | 125 | 136
  GHS/QoL Survival Follow-Up Month 6 | -2.00 [-6.16 to 2.16] | -3.37 [-7.24 to 0.50]
  GHS/QoL Survival Follow-Up Month 9: number analyzed (Participants) | 116 | 132
  GHS/QoL Survival Follow-Up Month 9 | -0.93 [-5.26 to 3.39] | -4.42 [-8.07 to -0.77]
  GHS/QoL Survival Follow-Up Month 12: number analyzed (Participants) | 111 | 126
  GHS/QoL Survival Follow-Up Month 12 | -1.65 [-5.91 to 2.61] | -4.50 [-8.67 to -0.32]
  GHS/QoL Survival Follow-Up Month 18: number analyzed (Participants) | 102 | 112
  GHS/QoL Survival Follow-Up Month 18 | -0.98 [-6.10 to 4.14] | -4.17 [-8.67 to 0.34]
  GHS/QoL Survival Follow-Up Month 24: number analyzed (Participants) | 83 | 108
  GHS/QoL Survival Follow-Up Month 24 | 1.31 [-3.50 to 6.12] | -6.17 [-10.96 to -1.39]
  GHS/QoL Survival Follow-Up Month 30: number analyzed (Participants) | 65 | 72
  GHS/QoL Survival Follow-Up Month 30 | -2.18 [-8.05 to 3.69] | -9.14 [-14.26 to -4.03]
  GHS/QoL Survival Follow-Up Month 36: number analyzed (Participants) | 62 | 69
  GHS/QoL Survival Follow-Up Month 36 | -1.08 [-6.42 to 4.27] | -5.56 [-11.22 to 0.11]
  GHS/QoL Survival Follow-Up Month 48: number analyzed (Participants) | 2 | 7
  GHS/QoL Survival Follow-Up Month 48 | -25.00 [-342.66 to 292.66] | -21.43 [-37.99 to -4.86]
  Physical Functioning Cycle 2 Day 1: number analyzed (Participants) | 163 | 157
  Physical Functioning Cycle 2 Day 1 | -6.37 [-8.58 to -4.16] | -5.73 [-8.18 to -3.29]
  Physical Functioning Cycle 3 Day 1: number analyzed (Participants) | 151 | 142
  Physical Functioning Cycle 3 Day 1 | -12.17 [-15.43 to -8.92] | -12.90 [-16.62 to -9.17]
  Physical Functioning Cycle 4 Day 1: number analyzed (Participants) | 151 | 149
  Physical Functioning Cycle 4 Day 1 | -19.48 [-22.51 to -16.45] | -21.68 [-25.66 to -17.70]
  Physical Functioning Cycle 5 Day 1: number analyzed (Participants) | 145 | 139
  Physical Functioning Cycle 5 Day 1 | -21.59 [-25.17 to -18.01] | -26.43 [-30.61 to -22.25]
  Physical Functioning Cycle 6 Day 1: number analyzed (Participants) | 134 | 132
  Physical Functioning Cycle 6 Day 1 | -10.20 [-13.46 to -6.94] | -12.20 [-15.39 to -9.00]
  Physical Functioning Cycle 7 Day 1: number analyzed (Participants) | 122 | 128
  Physical Functioning Cycle 7 Day 1 | -7.43 [-10.48 to -4.38] | -8.96 [-12.22 to -5.69]
  Physical Functioning Cycle 8 Day 1: number analyzed (Participants) | 119 | 122
  Physical Functioning Cycle 8 Day 1 | -4.80 [-7.52 to -2.09] | -7.70 [-11.21 to -4.19]
  Physical Functioning Cycle 9 Day 1: number analyzed (Participants) | 121 | 122
  Physical Functioning Cycle 9 Day 1 | -5.40 [-8.20 to -2.60] | -5.74 [-9.04 to -2.44]
  Physical Functioning Cycle 10 Day 1: number analyzed (Participants) | 114 | 122
  Physical Functioning Cycle 10 Day 1 | -4.87 [-7.82 to -1.92] | -6.17 [-9.25 to -3.10]
  Physical Functioning Cycle 11 Day 1: number analyzed (Participants) | 119 | 121
  Physical Functioning Cycle 11 Day 1 | -3.99 [-6.77 to -1.21] | -5.73 [-9.09 to -2.37]
  Physical Functioning Cycle 12 Day 1: number analyzed (Participants) | 119 | 122
  Physical Functioning Cycle 12 Day 1 | -2.59 [-5.39 to 0.21] | -6.61 [-9.60 to -3.62]
  Physical Functioning Cycle 13 Day 1: number analyzed (Participants) | 119 | 121
  Physical Functioning Cycle 13 Day 1 | -3.63 [-6.77 to -0.48] | -6.72 [-10.01 to -3.43]
  Physical Functioning Cycle 14 Day 1: number analyzed (Participants) | 119 | 117
  Physical Functioning Cycle 14 Day 1 | -3.42 [-6.33 to -0.51] | -5.07 [-8.25 to -1.89]
  Physical Functioning Cycle 15 Day 1: number analyzed (Participants) | 112 | 116
  Physical Functioning Cycle 15 Day 1 | -4.24 [-7.59 to -0.89] | -5.89 [-9.22 to -2.56]
  Physical Functioning Cycle 16 Day 1: number analyzed (Participants) | 111 | 114
  Physical Functioning Cycle 16 Day 1 | -2.42 [-5.70 to 0.86] | -5.79 [-9.05 to -2.53]
  Physical Functioning Study Drug Completion/Early Discontinuation: number analyzed (Participants) | 130 | 137
  Physical Functioning Study Drug Completion/Early Discontinuation | -5.58 [-8.88 to -2.27] | -8.66 [-12.12 to -5.21]
  Physical Functioning Survival Follow-Up Month 3: number analyzed (Participants) | 131 | 142
  Physical Functioning Survival Follow-Up Month 3 | -4.16 [-6.77 to -1.55] | -8.54 [-11.83 to -5.26]
  Physical Functioning Survival Follow-Up Month 6: number analyzed (Participants) | 125 | 136
  Physical Functioning Survival Follow-Up Month 6 | -5.21 [-7.90 to -2.53] | -6.91 [-10.10 to -3.72]
  Physical Functioning Survival Follow-Up Month 9: number analyzed (Participants) | 116 | 132
  Physical Functioning Survival Follow-Up Month 9 | -3.97 [-6.65 to -1.28] | -7.78 [-11.20 to -4.36]
  Physical Functioning Survival Follow-Up Month 12: number analyzed (Participants) | 111 | 126
  Physical Functioning Survival Follow-Up Month 12 | -4.43 [-7.23 to -1.62] | -7.46 [-11.07 to -3.85]
  Physical Functioning Survival Follow-Up Month 18: number analyzed (Participants) | 102 | 112
  Physical Functioning Survival Follow-Up Month 18 | -4.90 [-8.58 to -1.22] | -6.61 [-10.17 to -3.05]
  Physical Functioning Survival Follow-Up Month 24: number analyzed (Participants) | 82 | 108
  Physical Functioning Survival Follow-Up Month 24 | -4.07 [-7.64 to -0.49] | -6.30 [-9.94 to -2.65]
  Physical Functioning Survival Follow-Up Month 30: number analyzed (Participants) | 65 | 72
  Physical Functioning Survival Follow-Up Month 30 | -3.36 [-6.90 to 0.18] | -10.46 [-14.68 to -6.25]
  Physical Functioning Survival Follow-Up Month 36: number analyzed (Participants) | 62 | 69
  Physical Functioning Survival Follow-Up Month 36 | -4.06 [-8.93 to 0.81] | -8.70 [-12.47 to -4.92]
  Physical Functioning Survival Follow-Up Month 48: number analyzed (Participants) | 2 | 7
  Physical Functioning Survival Follow-Up Month 48 | -3.33 [-45.69 to 39.02] | -11.43 [-24.12 to 1.26]
  Role Functioning Cycle 2 Day 1: number analyzed (Participants) | 163 | 157
  Role Functioning Cycle 2 Day 1 | -8.08 [-12.05 to -4.11] | -12.42 [-16.70 to -8.14]
  Role Functioning Cycle 3 Day 1: number analyzed (Participants) | 151 | 142
  Role Functioning Cycle 3 Day 1 | -19.54 [-24.57 to -14.50] | -19.84 [-24.92 to -14.76]
  Role Functioning Cycle 4 Day 1: number analyzed (Participants) | 152 | 149
  Role Functioning Cycle 4 Day 1 | -28.29 [-33.49 to -23.09] | -33.56 [-39.19 to -27.93]
  Role Functioning Cycle 5 Day 1: number analyzed (Participants) | 145 | 139
  Role Functioning Cycle 5 Day 1 | -32.99 [-38.45 to -27.53] | -38.97 [-44.44 to -33.50]
  Role Functioning Cycle 6 Day 1: number analyzed (Participants) | 134 | 132
  Role Functioning Cycle 6 Day 1 | -22.39 [-27.55 to -17.23] | -26.14 [-31.45 to -20.83]
  Role Functioning Cycle 7 Day 1: number analyzed (Participants) | 122 | 128
  Role Functioning Cycle 7 Day 1 | -14.21 [-19.06 to -9.35] | -18.36 [-23.36 to -13.36]
  Role Functioning Cycle 8 Day 1: number analyzed (Participants) | 119 | 122
  Role Functioning Cycle 8 Day 1 | -10.50 [-15.16 to -5.85] | -14.89 [-20.37 to -9.41]
  Role Functioning Cycle 9 Day 1: number analyzed (Participants) | 121 | 122
  Role Functioning Cycle 9 Day 1 | -10.74 [-15.21 to -6.28] | -13.80 [-19.13 to -8.47]
  Role Functioning Cycle 10 Day 1: number analyzed (Participants) | 114 | 122
  Role Functioning Cycle 10 Day 1 | -9.36 [-13.94 to -4.77] | -13.39 [-18.13 to -8.64]
  Role Functioning Cycle 11 Day 1: number analyzed (Participants) | 119 | 122
  Role Functioning Cycle 11 Day 1 | -8.26 [-12.65 to -3.88] | -12.98 [-17.53 to -8.43]
  Role Functioning Cycle 12 Day 1: number analyzed (Participants) | 119 | 122
  Role Functioning Cycle 12 Day 1 | -6.86 [-11.40 to -2.33] | -13.52 [-18.06 to -8.99]
  Role Functioning Cycle 13 Day 1: number analyzed (Participants) | 119 | 121
  Role Functioning Cycle 13 Day 1 | -6.30 [-10.16 to -2.44] | -14.46 [-19.69 to -9.24]
  Role Functioning Cycle 14 Day 1: number analyzed (Participants) | 119 | 117
  Role Functioning Cycle 14 Day 1 | -7.28 [-11.77 to -2.80] | -13.82 [-18.80 to -8.84]
  Role Functioning Cycle 15 Day 1: number analyzed (Participants) | 112 | 116
  Role Functioning Cycle 15 Day 1 | -8.63 [-13.14 to -4.12] | -11.78 [-16.96 to -6.60]
  Role Functioning Cycle 16 Day 1: number analyzed (Participants) | 111 | 114
  Role Functioning Cycle 16 Day 1 | -4.65 [-9.70 to 0.39] | -10.82 [-15.56 to -6.07]
  Role Functioning Study Drug Completion/Early Discontinuation: number analyzed (Participants) | 130 | 137
  Role Functioning Study Drug Completion/Early Discontinuation | -8.46 [-13.54 to -3.38] | -16.42 [-21.64 to -11.21]
  Role Functioning Survival Follow-Up Month 3: number analyzed (Participants) | 131 | 142
  Role Functioning Survival Follow-Up Month 3 | -5.98 [-10.57 to -1.39] | -14.44 [-19.35 to -9.53]
  Role Functioning Survival Follow-Up Month 6: number analyzed (Participants) | 125 | 136
  Role Functioning Survival Follow-Up Month 6 | -10.67 [-15.66 to -5.68] | -13.97 [-18.84 to -9.10]
  Role Functioning Survival Follow-Up Month 9: number analyzed (Participants) | 116 | 132
  Role Functioning Survival Follow-Up Month 9 | -7.61 [-12.23 to -3.00] | -13.76 [-18.45 to -9.08]
  Role Functioning Survival Follow-Up Month 12: number analyzed (Participants) | 111 | 126
  Role Functioning Survival Follow-Up Month 12 | -7.66 [-11.90 to -3.41] | -12.83 [-18.13 to -7.53]
  Role Functioning Survival Follow-Up Month 18: number analyzed (Participants) | 102 | 112
  Role Functioning Survival Follow-Up Month 18 | -7.03 [-12.54 to -1.51] | -12.05 [-17.15 to -6.95]
  Role Functioning Survival Follow-Up Month 24: number analyzed (Participants) | 82 | 108
  Role Functioning Survival Follow-Up Month 24 | -9.96 [-15.85 to -4.07] | -10.96 [-16.19 to -5.72]
  Role Functioning Survival Follow-Up Month 30: number analyzed (Participants) | 65 | 72
  Role Functioning Survival Follow-Up Month 30 | -8.72 [-15.45 to -1.98] | -16.44 [-23.12 to -9.75]
  Role Functioning Survival Follow-Up Month 36: number analyzed (Participants) | 62 | 69
  Role Functioning Survival Follow-Up Month 36 | -5.65 [-12.45 to 1.16] | -12.56 [-18.94 to -6.18]
  Role Functioning Survival Follow-Up Month 48: number analyzed (Participants) | 2 | 7
  Role Functioning Survival Follow-Up Month 48 | -16.67 [-228.44 to 195.10] | -21.43 [-47.70 to 4.84]

11. Secondary Outcome: Percentage of Participants With at Least One Adverse Events (AEs)
Description: Percentage of participants with at least one adverse event.
Time Frame: From randomization and up to study final analysis data cut off on 28 September 2022.
Population: Safety population is defined as all participants who received any dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab and Chemotherapy | Placebo and Chemotherapy
Number analyzed (Participants) | 164 | 167
Percentage of participants | 100 | 100

12. Secondary Outcome: Minimum Observed Serum Atezolizumab Concentration (Cmin)
Description: Minimum observed serum atezolizumab concentration.
Time Frame: Pre-dose on Day 1 of Cycles 2, 3, 4, 6, 8, 12, and 16 (cycle length = 28 days from Cycles 1 to 5, and 21 days from Cycles 6 to 16)
Population: The pharmacokinetic-evaluable population is defined as all participants who received any dose of atezolizumab and who have evaluable pharmacokinetic (PK) samples.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 164
µg/mL
  Cycle 2 Day 1 | 142 (54.3)
  Cycle 3 Day 1 | 189 (64.2)
  Cycle 4 Day 1 | 207 (77.3)
  Cycle 6 Day 1 | 78.7 (50.3)
  Cycle 8 Day 1 | 204 (62.7)
  Cycle 12 Day 1 | 267 (81.1)
  Cycle 16 Day 1 | 303 (89.1)

13. Secondary Outcome: Maximum Observed Serum Atezolizumab Concentration (Cmax)
Description: Maximum observed atezolizumab concentration (Cmax).
Time Frame: Day 1 of Cycle 1 post dose (cycle length = 28 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 164
µg/mL | 334 (63.3)

14. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: Percentage of participants with anti-drug antibodies (ADAs) to atezolizumab.
Time Frame: Baseline up to approximately 20 months
Population: The anti-drug antibodies (ADA)-evaluable population is defined as all participants treated with atezolizumab who have at least one post-baseline ADA result.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 162
Percentage of participants
  Baseline evaluable participants | 2.5
  Post-baseline evaluable participants: number analyzed (Participants) | 157
  Post-baseline evaluable participants | 13.4

ADVERSE EVENTS:
Time Frame: From the first study drug and up to study final analysis data cut off on 28 September 2022, up to approximately 62 months.
Description: Safety population included participants who received any amount of any study drug.
Arm/Group | Placebo and Chemotherapy | Atezolizumab and Chemotherapy
All-Cause Mortality (participants affected / at risk) | 28/167 | 16/164
Serious Adverse Events (participants affected / at risk) | 36/167 | 59/164
Other Adverse Events (participants affected / at risk) | 167/167 | 162/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Chemotherapy (N=167) | Atezolizumab and Chemotherapy (N=164)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (14) | 16 (18)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bacillus bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Chemotherapy (N=167) | Atezolizumab and Chemotherapy (N=164)
Anaemia (Blood and lymphatic system disorders) | 65 (80) | 64 (89)
Leukopenia (Blood and lymphatic system disorders) | 17 (29) | 23 (46)
Neutropenia (Blood and lymphatic system disorders) | 59 (123) | 65 (141)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 13 (16)
Hypothyroidism (Endocrine disorders) | 0 (0) | 22 (22)
Dry eye (Eye disorders) | 6 (6) | 13 (13)
Lacrimation increased (Eye disorders) | 18 (18) | 18 (21)
Vision blurred (Eye disorders) | 11 (12) | 16 (16)
Abdominal pain (Gastrointestinal disorders) | 16 (21) | 23 (29)
Abdominal pain upper (Gastrointestinal disorders) | 13 (16) | 21 (23)
Constipation (Gastrointestinal disorders) | 55 (64) | 51 (74)
Diarrhoea (Gastrointestinal disorders) | 74 (117) | 74 (110)
Dry mouth (Gastrointestinal disorders) | 5 (6) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 21 (23) | 19 (22)
Nausea (Gastrointestinal disorders) | 110 (189) | 108 (218)
Stomatitis (Gastrointestinal disorders) | 29 (32) | 40 (48)
Vomiting (Gastrointestinal disorders) | 51 (70) | 63 (105)
Asthenia (General disorders) | 36 (40) | 42 (66)
Fatigue (General disorders) | 65 (86) | 65 (94)
Malaise (General disorders) | 17 (18) | 15 (35)
Mucosal inflammation (General disorders) | 15 (19) | 18 (24)
Oedema peripheral (General disorders) | 24 (27) | 24 (30)
Pain (General disorders) | 11 (11) | 20 (22)
Pyrexia (General disorders) | 21 (25) | 37 (55)
Nasopharyngitis (Infections and infestations) | 14 (17) | 23 (29)
Paronychia (Infections and infestations) | 21 (21) | 19 (20)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 23 (30)
Urinary tract infection (Infections and infestations) | 11 (11) | 18 (25)
Infusion related reaction (Injury, poisoning and procedural complications) | 10 (16) | 16 (28)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 14 (17)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 32 (32)
Alanine aminotransferase increased (Investigations) | 35 (53) | 39 (63)
Aspartate aminotransferase increased (Investigations) | 28 (44) | 37 (64)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 14 (19)
Blood lactate dehydrogenase increased (Investigations) | 7 (7) | 10 (11)
Neutrophil count decreased (Investigations) | 30 (67) | 29 (60)
Weight decreased (Investigations) | 8 (8) | 15 (17)
White blood cell count decreased (Investigations) | 15 (35) | 14 (33)
Decreased appetite (Metabolism and nutrition disorders) | 33 (36) | 28 (37)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (9) | 12 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (61) | 50 (76)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (24) | 24 (27)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 13 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 40 (49) | 51 (86)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (26) | 27 (36)
Dizziness (Nervous system disorders) | 15 (16) | 20 (33)
Dysgeusia (Nervous system disorders) | 25 (27) | 16 (20)
Headache (Nervous system disorders) | 36 (46) | 51 (86)
Neuropathy peripheral (Nervous system disorders) | 34 (42) | 40 (48)
Paraesthesia (Nervous system disorders) | 19 (22) | 12 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 42 (45) | 58 (65)
Polyneuropathy (Nervous system disorders) | 14 (15) | 10 (10)
Taste disorder (Nervous system disorders) | 13 (13) | 10 (11)
Anxiety (Psychiatric disorders) | 11 (11) | 12 (13)
Depression (Psychiatric disorders) | 6 (6) | 11 (11)
Insomnia (Psychiatric disorders) | 29 (30) | 49 (61)
Breast pain (Reproductive system and breast disorders) | 15 (15) | 17 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (39) | 41 (52)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 23 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 25 (26)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 19 (20)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 129 (132) | 125 (127)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 (10) | 6 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (13) | 18 (20)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 15 (17)
Nail discolouration (Skin and subcutaneous tissue disorders) | 29 (29) | 26 (28)
Nail disorder (Skin and subcutaneous tissue disorders) | 10 (10) | 21 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (31) | 36 (49)
Rash (Skin and subcutaneous tissue disorders) | 42 (53) | 52 (68)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (14) | 12 (12)
Hot flush (Vascular disorders) | 17 (20) | 28 (32)
Hypertension (Vascular disorders) | 17 (29) | 15 (27)

LIMITATIONS AND CAVEATS:
This study was not designed nor formally powered to demonstrate statistically significant improvements in the secondary efficacy endpoints of EFS, DFS and OS. The analyses of these secondary endpoints are descriptive in nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT03197935/Prot_002.pdf
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT03197935/SAP_001.pdf